CLINICAL TRIAL: NCT01227733
Title: Comparative Genomic and Genetic Analysis of Paired Primary Breast - Metastatic Tumor Specimens Using High-throughput Platforms
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: National University Hospital, Singapore (Other)
Other Study IDs: BR06/25/10
Record Dates: First submitted 2010-10-21; First posted 2010-10-25 (Estimated); Last update posted 2014-01-22 (Estimated); Status verified 2014-01

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Breast Tumor: Breast Tumor Blocks
  Interventions: Other: Breast Tumor Blocks

INTERVENTIONS:
Other: Breast Tumor Blocks

SUMMARY:
Adequate quality and quantity of RNA may be extracted from paraffin-embedded tumor blocks for gene expression analysis. This has clinical relevance as gene expression signatures may then be profiled using archival tumor blocks, which are more readily available than frozen tissues.

ELIGIBILITY:
Inclusion Criteria:

No participants are involved.

Exclusion Criteria:

No participants are involved.

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Up to 10 archival breast tumor blocks will be obtained from the Department of Pathology, NUH - half of these blocks will be from patients who were diagnosed before year 2000, and the other half of the blocks will be from patients diagnosed between year 2000-2005 (control specimens). Basic tumor and patient information will be collected without patient identifiers - grade, stage, ER/PR/HER2 status, treatment received, outcome data. 8-10 ten-micron sections will be cut from each tumor block. RNA will be extracted from the tumor sections using the Roche High Pure FFPE RNA Micro Kit. RNA will be profiled using the Illumina Veracode assay and the Affymetrix Quantigene assay. RNA extraction and gene expression profiling will be performed by collabroators at the Genome Institute of Singapore.
Sampling Method: Non-Probability Sample
Dates: Start 2010-08; Primary Completion 2014-12 (Estimated); Study Completion 2014-12 (Estimated)

CONTACTS AND LOCATIONS:
Locations (1):
- National University Hospital, Singapore, Singapore, Singapore

REFERENCES:
- [Background] Barrios CH, Liu MC, Lee SC, Vanlemmens L, Ferrero JM, Tabei T, Pivot X, Iwata H, Aogi K, Lugo-Quintana R, Harbeck N, Brickman MJ, Zhang K, Kern KA, Martin M. Phase III randomized trial of sunitinib versus capecitabine in patients with previously treated HER2-negative advanced breast cancer. Breast Cancer Res Treat. 2010 May;121(1):121-31. doi: 10.1007/s10549-010-0788-0. Epub 2010 Mar 26. PMID 20339913
- [Background] Lim YW, Goh BC, Wang LZ, Tan SH, Chuah BYS, Lim SE, Iau P, Buhari SA, Chan CW, Sukri NB, Cordero MT, Soo R, Lee SC. Pharmacokinetics and pharmacodynamics of docetaxel with or without ketoconazole modulation in chemonaive breast cancer patients. Ann Oncol. 2010 Nov;21(11):2175-2182. doi: 10.1093/annonc/mdq230. Epub 2010 Apr 29. PMID 20430905